CLINICAL TRIAL: NCT06187766
Title: Effects of Social Media Addiction on Physical Activity Level and Exercise Capacity in University Students
Status: Active, not recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Assistant Professor, Gazi University
Other Study IDs: 220819
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Addiction; Social Media Addiction; Physical Inactivity
MeSH Terms: conditions — Behavior, Addictive; Internet Addiction Disorder; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University Students: University students will be categorized with Bergen Social Media Addiction Scale.
  Interventions: Diagnostic Test: Social Media Addiction

INTERVENTIONS:
Diagnostic Test: Social Media Addiction — Social Media Addiction level will be determined by Bergen Social Media Addiction Scale

SUMMARY:
The aim of this study is to investigate the effect of social media addiction on functional exercise capacity and maximal exercise capacity in university students.

DETAILED DESCRIPTION:
The internet, one of the new communication technologies, has become an indispensable part of human life as it makes people's lives easier, provides people with the advantage of saving time, and facilitates and accelerates information acquisition.

Thanks to the internet, people can do many daily tasks quickly with minimal physical effort and cost. This makes personal and business life easier. Internet technology has many positive features. This network, which develops and changes daily, has become indispensable for many people. In addition to all these positive features, today, this situation emerges as a new addiction phenomenon. In cases where there is no parental or teacher supervision in their use of social media, adolescents encounter negative content.

There is a high probability of being affected by the contents. Sharing sites such as Facebook, Instagram, Twitter, Linkedin, YouTube, and Tumblr, which are very popular social media networks that have entered our lives, have been used by many people in the world and in Turkey for a long time. It seems that the rapid increase in usage rates and durations will continue rather than decrease.

The intense amount and duration of use brings the phenomenon of "addiction" to the agenda. People seek and express in virtual environments what they cannot achieve or express freely in real life. These types of actions increase people's usage time, So much so that this situation causes addiction. Many studies have been conducted in the literature to investigate the effect of social media and digital game addiction on physical activity levels. Although many studies have been conducted to examine social media addiction and the effects it causes, there is no research on the effects of social media addiction on functional exercise capacity and maximal exercise capacity. No study has been found investigating its effect. For this reason, the investigators think that there is a need for a study in this direction in the literature. The aim of this study is to investigate the effect of social media addiction on functional exercise capacity and maximal exercise capacity in university students.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-30 years

Exclusion Criteria:

* chronic illnesses
* can't walk or run

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Social Media Addiction | Baseline
  Bergen Social Media Addiction Scale is a social media addiction scale, but social media has been defined as the use of Facebook, Twitter, Instagram, etc. Therefore, BSMAS can be considered a SNA scale despite being called a social media addiction scale. BSMAS is an adaptation of Bergen Facebook addiction scale (BFAS). In BSMAS, the term "Facebook" has been replaced with "Social media" in all items of the scale. There is one item each for six components of behavioral addiction.Higher scores mean a social media addiction level is high.
Physical Activity Level | Baseline
  Physical activity will be evaluated using the International Physical Activity Questionnaire Short Form (IPAQ-SF), whose reliability and validity are documented . The questionnaire referre to the last 7 days and asked about walking, moderate-intensity activities, vigorous-intensity activities and sitting time.
Functional exercise capacity | Baseline
  The 6-min walk test (6MWT) will perform in a 30-m unobstructed corridor. Measurement will be done according to American Thoracic Society guidelines.
Maximal exercise capacity | Baseline
  A modified incremental shuttle walk test will be used to evaluate maximal exercise capacity.Subjects will be instructed to walk/run up and down a 10-m course marked by cones placed 0.5 m from each end.

CONTACTS AND LOCATIONS:
Overall Officials: Muserrefe Nur Keles, PhD, Study Chair — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation Recruiting Ankara, Turkey, 06500, Ankara, Turkey (Türkiye)